CLINICAL TRIAL: NCT06278571
Title: Efecto de la educación a través de Una aplicación móvil Con Reforzamiento médico y Nutricional Para Incidir en el Control metabólico, Conocimientos y Estilo de Vida de Los Pacientes Con Diabetes Tipo 2
Brief Title: Effect of Education With Mobile App on Metabolic Control in Patients With Type 2 Diabetes
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Coordinación de Investigación en Salud, Mexico (Other Government)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: R-2018-785-100
Record Dates: First submitted 2024-02-16; First posted 2024-02-26 (Actual); Last update posted 2025-04-24 (Actual); Status verified 2025-01

CONDITIONS: Female
MeSH Terms: interventions — Amyloid; Control Groups; Nutrition Therapy

STUDY DESIGN:
Intervention Model Description: Multicenter clinical trial
Who Masked: Participant
Masking Description: Participants are unaware of other intervention arms
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Intervention with mobile application and website (Experimental): Group with educational site and mobile App
  Interventions: Behavioral: Educational intervention with App and web site education; Behavioral: Educational interventión with web site education
- Group with educational site (Active Comparator): Group with educational site
  Interventions: Behavioral: Educational interventión with web site education; Other: Control group with nutritional therapy
- Control Group (No Intervention): Group with the usual care

INTERVENTIONS:
Behavioral: Educational intervention with App and web site education — This group will only receive intervention with access to the educational website from home, where they will review the different modules focused on diabetes care, nutrition and exercise. in addition to the usual medical care by your treating physician.
  Arms: Intervention with mobile application and website
Behavioral: Educational interventión with web site education — This group will receive, in addition to nutritional therapy, diabetes education through an educational site, to learn more about the most important aspects of diabetes care. In addition to the usual medical care by your treating physician.
  Arms: Group with educational site; Intervention with mobile application and website
Other: Control group with nutritional therapy — This group will receive only the usual medical care by your treating physician.
  Arms: Group with educational site

SUMMARY:
The objective of this study is to compare the effect of education through a mobile application with medical and nutritional reinforcement on the metabolic control of Mexican patients with type 2 diabetes attending primary care clinics in Mexico.

The research question is: What is the effect of education through a mobile application with medical and nutritional reinforcement vs.

nutritional and medical reinforcement, versus an educational platform to influence the metabolic control of patients with type 2 diabetes? Multicenter clinical trial in six family medicine units of the Mexican Institute of Social Security. These selected units are: UMF 9, UMF 28, UMF 7, UMF 1, UMF 9 and UMF 10.

Patients with type 2 diabetes will be randomly assigned to the educational intervention through the educational site, (n=160 patients), two clinics will be assigned for the use of the mobile App and the educational site (n=160 patients), and two clinics will be part of the control group (n=160 patients).

DETAILED DESCRIPTION:
Groups with educational website Participants will be invited to review the site at least once a week. There will be access to social networks and experts' blog for interaction with the patient, as well as an email for doubts with the researchers. The educational site has different educational modules that the patient can review dynamically, reinforcement messages and didactic activities at the end of each module to reinforce the learning acquired. The user will have free access to the educational platform. The educational site will automatically record the number of visits, modules and date of review and will be stored in a database. The above in order to measure adherence to the educational platform.

Groups with educational site and App for reinforcement This group will have access to the App-DM2, which will be installed on the cell phones of patients with diabetes, will have a record for a family member who will serve as a support network for the review of the APP-DM2. It will be compatible with the Android platform. At the beginning of the study the researchers will register each patient and they will receive via SMS message and/or email. The software will be compatible with both Android Smartphone. The investigator will ask the patient to download the application for their initial visit and review it on subsequent visits.

The control group will receive personalized counseling at the beginning of the study, both medical and nutritional, and will continue with their usual medical treatment provided in their family medicine units.

All patients will be scheduled at 3, 6 and 12 months of follow-up for capillary glucose, blood pressure, anthropometry and body composition measurements as follow-up and monitoring measures. In all patients at baseline, 6 and 12 months, venous blood biochemical, clinical, anthropometric and dietary variables will be measured and used for statistical analysis.

ELIGIBILITY:
Inclusion criteria

* Patients with type 2 diabetes.
* Enrolled as beneficiaries of the Mexican Social Security Institute.
* With HbA1 greater than 7% and less than 13%.
* With and without pharmacological treatment for diabetes (hypoglycemic agents or insulin).
* Who can read and write.
* With ≤ 60 years of age7.
* With ≤10 years of diabetes diagnosis.

Exclusion criteria

* chronic kidney disease with renal replacement therapy
* blindness
* lower limb amputation
* cancer

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 480 (Actual)
Dates: Start 2023-01-30 (Actual); Primary Completion 2025-04-30 (Estimated); Study Completion 2025-09-03 (Estimated)

PRIMARY OUTCOMES:
Number of participants with glycosylated hemoglobin at control goals | 12 months
  Glycosylated hemoglobin
Number of participants with iipid profile in control targets | The baseline and 12 months after the intervention will be evaluated.
  Assessment of the effect of the intervention on lipid profile
Number of participants with body mass index profile in control target | The baseline and 12 months after the intervention will be evaluated.
  Weight and height will be measured at baseline and at 12 months to obtain the body mass index.

SECONDARY OUTCOMES:
Number of patients with changes to a healthy lifestyle | The baseline and 12 months after the intervention will be evaluated.
  Lifestyle will be measured at baseline and 12 months through a validated questionnaire.
The proportion of patients with adequate knowledge of diabetes | The baseline and 12 months after the intervention will be evaluated.
  The proportion of patients with adequate knowledge of diabetes will be measured at baseline and 12 months.

CONTACTS AND LOCATIONS:
Overall Officials: Lubia Velazquez, PhD, Principal Investigator — UIEC. HGR 1. IMSS
Locations (1):
- Instituto Mexicano Del Seguro Social, Mexico City, Mexico City, Mexico

REFERENCES:
- [Derived] Torres San Miguel GP, Sevilla Gonzalez ML, Lopez Ramirez E, Flores Lopez MF, Velazquez Lopez L. Effect of a Mediterranean Diet Adapted to the Mexican Population on Indicators of Metabolic Risk in Patients With Obstructive Sleep Apnea: Protocol for a Randomized Controlled Trial. JMIR Res Protoc. 2025 Aug 21;14:e72513. doi: 10.2196/72513. PMID 40839868